CLINICAL TRIAL: NCT02844634
Title: Use of Tenofovir/Emtricitabine With Immediate or Deferred Doxycycline 100mg PO Daily for Combination HIV and Syphilis Pre-exposure Prophylaxis in HIV-negative Men Who Have Sex With Men: a Pilot Study of Dual Daily HIV and Syphilis PrEP. (The DuDHS Trial).
Brief Title: Tenofovir/Emtricitabine With Doxycycline for Combination HIV and Syphilis Pre-exposure Prophylaxis in HIV-negative MSM
Acronym: DuDHS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: British Columbia Centre for Disease Control (Other Government)
Responsible Party: Principal Investigator, Jonathan Troy Grennan, Physician Lead HIV/STI Program, British Columbia Centre for Disease Control
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BritishCCDC
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: HIV; Syphilis
Keywords: pre-exposure prophylaxis; men who have sex with men; HIV prevention; sexually transmitted infection; syphilis
MeSH Terms: conditions — Syphilis; Homosexuality; Sexually Transmitted Diseases | interventions — Doxycycline; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate doxycycline 100mg PO daily (Experimental): Individuals will receive tenofovir/emtricitabine one tablet daily in an open-label fashion.
  Subjects are randomized to immediate (12 months duration) doxycycline 100mg PO daily.
  Interventions: Drug: Doxycycline 100mg PO daily x 12 months; Drug: Tenofovir/emtricitabine 200/300mg PO daily
- Deferred doxycycline 100mg PO daily (Active Comparator): Individuals will receive daily tenofovir/emtricitabine one tablet daily and will begin doxycycline 100mg PO daily after 6 months for a total duration of 6 months
  Interventions: Drug: Tenofovir/emtricitabine 200/300mg PO daily; Drug: Doxycycline 100mg PO daily x 6 months

INTERVENTIONS:
Drug: Doxycycline 100mg PO daily x 12 months — Immediate use of daily doxycycline (12 months duration, to start immediately)
  Arms: Immediate doxycycline 100mg PO daily
Drug: Tenofovir/emtricitabine 200/300mg PO daily — Daily use of tenofovir/emtricitabine
Drug: Doxycycline 100mg PO daily x 6 months — Deferred use of doxycycline (6 months duration, to start 6 months post-randomization)
  Arms: Deferred doxycycline 100mg PO daily

SUMMARY:
Men who have sex with men remain at high risk for HIV infection. Targeting prevention interventions to MSM at highest risk of seroconversion is an important goal of combination prevention interventions. Antecedent diagnosis of another sexually transmitted infection (STI), particularly syphilis, may serve as an entry point for biomedical prevention as these individuals are at highest risk for incident HIV. The use of the antiretroviral combination of tenofovir/emtricitabine has been shown to be associated with an overall 44% reduction in HIV acquisition in high-risk MSM when taken daily as PrEP. In those individuals with detectable drug levels, the benefit was as high as 90% risk reduction. In real-world evaluations of PrEP, high-risk sexual behaviour may continue as evidenced by high rates of intercurrent sexually transmitted infections. As such, biomedical interventions that may offer additional reduction in acquisition of common sexually transmitted infections should also be evaluated.

Recently a small pilot study has demonstrated potential benefit from a similar strategy for syphilis prevention. In this study 30 MSM were randomized to receive either 100mg doxycycline once daily or contingency management strategies linked to remaining free of sexually transmitted diseases at progressive study visits. Overall, those receiving doxycycline were significantly less likely to be diagnosed with any STI during followup than those in the comparator arm.

The investigators therefore propose to undertake a pilot study to evaluate the feasibility of using both tenofovir/emtricitabine and doxycycline (immediate or deferred use) for pre-exposure prophylaxis amongst HIV-negative MSM with recent history of syphilis infection in Vancouver, Canada.

DETAILED DESCRIPTION:
1. Rationale:

   1.1 Men who have sex with men with antecedent diagnosis of another sexually transmitted infection, particularly syphilis, are at high risk for HIV infection.

   Men who have sex with men (MSM) continue to experience high rates of HIV incident infections in Canada and a disproportionately high burden of disease relative to the general population. In 2011, approximately 48% of new diagnoses occurred in MSM across Canada, a figure that has been relatively stable for the last decade. Within British Columbia (BC), although HIV new diagnosis rates overall have been declining over the last decade (dropping from a rate of 10.6 cases/100,000 in 2004 to 5.9 cases/100,000 in 2013), MSM made up an increasing majority of new diagnoses (59%) within BC in 2013. Within Vancouver Coastal Health Authority (VCH), approximately 70% of all new HIV diagnoses annually from 2012-15 were amongst MSM.

   Targeting prevention interventions to MSM at highest risk is important when determining potential publicly funded biomedical interventions, particularly the use of HIV pre-exposure prophylaxis (PrEP). Antecedent diagnosis of another sexually transmitted infection (STI) may serve as an entry point for biomedical prevention as these individuals are at highest risk for incident HIV. In an evaluation of HIV incidence following diagnosis of syphilis infection in New York City, the annual HIV incidence was 3.6% (95% Confidence Interval [CI]: 3.27% - 3.97%), with overall HIV incidence amongst MSM of 5.56% (1). In those males with syphilis and a subsequent additional STI the HIV incidence was even greater at 7.89% (95% CI: 6.62% - 9.24%). A similar analysis of clients attending STI clinics in BC has revealed that antecedent STI is predictive of an elevated risk for subsequent HIV seroconversion with clients who ever had a diagnosis of syphilis having an HIV incidence of 3.6% person-years (95%CI: 2.5-4.9), gonorrhea (2.0%; 95%CI: 1.6-2.5), rectal gonorrhea (4.5% person-years; 95%CI: 3.4-5.8), while individuals with rectal gonorrhea and syphilis had an incidence rate of 12.6 % person-years (95%CI: 8.4-21.8).

   Evaluating the use of PrEP in MSM with antecedent STI is an important component to inform HIV prevention programs in BC and nationally. The STI clinics operated by the BC Centre for Disease Control are well-positioned for this evaluation as about 15 and 25% of all HIV diagnoses in BC and VCH, respectively are diagnosed at these clinics.

   1.2. STI prevention strategies may also benefit from biomedical prevention interventions

   Novel biomedical strategies have been shown to be effective in preventing acquisition of STI such as HIV, and are now considered to be standard of care for at-risk MSM in the United States. The use of the antiretroviral combination of tenofovir/emtricitabine has been shown to be associated with an overall 44% reduction in HIV acquisition in high-risk MSM when taken daily as PrEP. In those individuals with detectable drug levels, the benefit was as high as 90% risk reduction. In real-world evaluations of PrEP, high-risk sexual behaviour may continue as evidenced by high rates of intercurrent STI (50% of PrEP users after 12 months in a study of 657 PrEP initiators in San Francisco). As such, biomedical interventions that may offer additional reduction in acquisition of common sexually transmitted infections should be evaluated.

   Recently a small pilot study has demonstrated potential benefit from a similar strategy for syphilis prevention (2). In this study 30 MSM were randomized to receive either 100mg doxycycline once daily or contingency management strategies linked to remaining free of sexually transmitted diseases at progressive study visits. Doxycycline 100mg daily was chosen based on prior studies indicating that doses as low as once weekly doxycycyline could serve as prophylaxis for leptospirosis, another spirochete infection.

   Overall, those receiving doxycycline were significantly less likely to be diagnosed with any STI during follow-up than those in the comparator arm (odds ratio [OR] 0.27; 95% CI 0.09 - 0.83). Specific protection against syphilis infection was not seen during the on-treatment phase (OR 0.27; 95% CI 0.04 - 1.73), possibly reflecting the small sample size. During the study period, no change in sexual behaviours between arms was noted, supporting the potential role of doxycycline prophylaxis. A larger pilot evaluation of this strategy, in combination with HIV PrEP, would be a novel syndemic approach to addressing both the HIV and syphilis burden amongst the highest risk MSM.

   The investigators therefore propose to undertake a randomized trial of immediate vs. deferred doxycycline in conjunction with daily tenofovir/emtricitabine to determine the feasibility of combined HIV and syphilis pre-exposure prophylaxis amongst HIV-negative MSM with recent history of syphilis infection in Vancouver, Canada.
2. Objectives:

We propose to undertake a pilot trial of immediate vs. deferred doxycycline in conjunction with daily tenofovir/emtricitabine to determine the feasibility of combined HIV and syphilis pre-exposure prophylaxis amongst HIV-negative MSM with recent history of syphilis infection in Vancouver, Canada. We will meet this aim through the following objectives:

1. To assess feasibility of using dual daily HIV and syphilis PrEP, as defined by:

   a. Evaluation of feasibility of recruitment for a larger study i. Proportion of participants approached for study who are eligible and agree to participate.

   b. Adherence to 6 or 12 months of tenofovir/emtricitabine and doxycycline i. Determine proportion of individuals with >95% adherence to dual therapy over 6 and 12 months ii. Proportion of individuals with detectable doxycycline plasma level at each study visit.

   Additional measures of feasibility will include the assessment of:

   c. Tolerability of dual PrEP i. Comparison of grade 3 or 4 adverse events in those receiving immediate vs. deferred PrEP
2. To evaluate antimicrobial resistance over time.

   a. Change in proportion of participants with evidence of tetracycline class resistance in common flora, namely Staphylococcus aureus, Streptococcus pyogenes and Streptococcus pneumoniae from baseline to 6 and 12 months.

   Secondary objectives will include:
3. To evaluate changes in sexual activity reported by study participants over the study period.
4. To compare syphilis incidence between those in the immediate vs. deferred doxycycline arms.
5. To describe frequency of other STI's diagnosed in study participants over the study period.

   Exploratory objectives will include:
6. To evaluate doxycycline resistance in individuals with documented T.pallidum infection.
7. To evaluate HIV incidence and syphilis re-infection rates over a 12 month period.
8. Characterize changes in the rectal microbiome from baseline to 6 and 12 months after initiation of doxycycline

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years of age.
2. Self-reported MSM status.
3. Self-report condomless anal sex with a man within the last 6 months.
4. HIV negative based on HIV nucleic acid amplification testing (NAT).
5. Prior diagnosis of syphilis within preceding 36 months (defined on the basis of a new positive serum rapid plasma reagin (RPR) test, or ≥2-dilution rise in titre if previous syphilis, or positive darkfield microscopy result or T. pallidum direct fluorescent antibody test or PCR from a primary lesion).
6. Able to provide informed consent.

Exclusion Criteria:

1. HIV-positive individuals.
2. Recent (within last 30 days) use of HIV post-exposure prophylaxis (PEP).
3. Impaired renal function defined as glomerular filtration rate < 60 mL/min.
4. Chronic active Hepatitis B infection.
5. History of myasthenia gravis.
6. History of tetracycline/doxycycline allergy.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who are eligible and consent to participate amongst those approached. | 12 months
  To evaluate the feasibility of recruitment for a larger study
Proportion of participants reporting > 95% adherence to both HIV and syphilis PrEP therapies | 12 months
  To assess adherence of dual HIV and syphilis PrEP therapies
The proportion of individuals with detectable doxycycline at each study time point. | 12 months
  To assess adherence of syphilis PrEP therapy
The proportion of individuals reporting grade 3 or 4 adverse events in the immediate vs. deferred arms. | 12 months
  To assess the tolerability of dual HIV and syphilis PrEP therapies
The proportion of individuals with evidence of tetracycyline class resistance in common flora | 6 and 12 months
  To evaluate antimicrobial resistance over time

SECONDARY OUTCOMES:
To evaluate changes in sexual activity reported by study participants over the study period. | 12 months
  Evaluation of sexual activity over time
To evaluate incidence of recurrent syphilis re-infection stratified by use immediate versus deferred doxycycline PrEP. | 12 months
  Evaluation of syphilis incidence rates between the two study arms
To describe incidence of gonorrhea or chlamydia infection over the study period. | 12 months
  Assessment of the frequency of other STIs over time

OTHER OUTCOMES:
To assess the incidence of HIV in study participants | 12 months
  Exploratory outcome to access incidence rates for HIV infection
To assess the incidence of doxycycline resistance in those with documented T. pallidum infection. | 12 months
  Exploratory outcome to assess incidence rates for doxycycline resistance
To assess the changes in the composition of the rectal microbiome | 6 and 12 months
  Exploratory outcome to determine percentage changes in the bacterial genius of the rectal microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Troy Grennan, MD, Principal Investigator — BC Centre for Disease Control
Locations (1):
- BC Centre for Disease Control, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pathela P, Braunstein SL, Blank S, Shepard C, Schillinger JA. The high risk of an HIV diagnosis following a diagnosis of syphilis: a population-level analysis of New York City men. Clin Infect Dis. 2015 Jul 15;61(2):281-7. doi: 10.1093/cid/civ289. Epub 2015 Apr 13. PMID 25870333
- [Result] Bolan RK, Beymer MR, Weiss RE, Flynn RP, Leibowitz AA, Klausner JD. Doxycycline prophylaxis to reduce incident syphilis among HIV-infected men who have sex with men who continue to engage in high-risk sex: a randomized, controlled pilot study. Sex Transm Dis. 2015 Feb;42(2):98-103. doi: 10.1097/OLQ.0000000000000216. PMID 25585069